CLINICAL TRIAL: NCT06966557
Title: Treatment of Chronic Temporomandibular Pain With Peripheral Nerve Block
Brief Title: Nerve Block Treatment for Chronic Jaw Pain
Status: Recruiting | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: BnaiZion -TMJ2025
Record Dates: First submitted 2025-05-04; First posted 2025-05-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: TMJ Pain
Keywords: TMJ Pain; Nerve block; Peripheral nerve block; Chronic temporomandibular pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Study Summary: Nerve Block Treatment for Chronic Jaw Pain This study is being conducted at the TMJ (temporomandibular joint) clinic, which is part of the oral and maxillofacial surgery department. The goal is to evaluate how effective peripheral nerve blocks are in reducing long-term jaw pain in patients with chronic temporomandibular disorders (TMD) who haven't responded to at least two other types of treatment (such as physical therapy, medication, or bite splints).

What Is the Treatment? Peripheral nerve blocks are injections that temporarily block nerve signals from the painful area. This can relieve pain and improve function. These blocks are already used routinely at the clinic.

Who Can Join? Adults who have had jaw joint pain for over a year.

Have tried at least two other treatments without success.

Are mentally competent and not pregnant.

What Will Participation Involve? You'll receive the nerve block treatment as part of your regular care.

You'll be asked to attend follow-up visits, typically one every 4 months (3 per year).

You'll be monitored for pain relief, mouth opening ability, and use of pain medications.

You can stop participating at any time without affecting your care.

How Will Data Be Handled? Your information will be stored securely and coded to protect your identity.

Only the research team will have access to your personal information.

How Many People Will Be in the Study? The goal is to recruit 40 patients.

DETAILED DESCRIPTION:
Background:

Chronic temporomandibular disorders (TMD) are a common source of orofacial pain, affecting both younger and older populations. Symptoms often include sharp, persistent pain in the temporomandibular joint (TMJ) region, difficulty opening or closing the mouth, and functional limitations in the jaw and facial muscles. The condition may arise from various causes, including trauma, genetic predisposition, and muscular or joint stress.

Conventional treatments-such as medications, physiotherapy, bite splints, and complementary therapies-offer relief to many patients, but a subset remains resistant to these modalities. In recent years, peripheral nerve blocks have emerged as a promising intervention for managing chronic TMD-related pain, particularly in patients unresponsive to standard care.

Purpose of the Study:

This prospective observational study aims to systematically assess the effectiveness of peripheral nerve blocks as a treatment for chronic temporomandibular pain. The intervention is already part of routine clinical care in the TMJ clinic, and this study will evaluate patient outcomes in a structured manner.

Study Design and Methods:

Patients attending the TMJ clinic at our institution, who meet specific inclusion criteria, will be invited to participate in a follow-up study after receiving a peripheral nerve block as part of their clinical care. The treatment involves injecting anesthetic near specific nerves to block pain signals from the TMJ region.

Data will be collected prospectively from up to 40 adult participants. Baseline and follow-up data will include:

Pain levels (using the Visual Analog Scale - VAS)

Mouth opening range (in millimeters)

Changes in the use of pain medication

Whether the patient requests repeat treatments

Demographics and relevant medical background (age, sex, comorbidities, previous treatments, physical activity)

Follow-up visits will occur as per the clinic's standard practice, typically every four months (total of three visits per year), with the possibility for earlier visits if symptoms worsen. Patients must attend at least two follow-up visits within four months post-injection to remain in the study.

Inclusion Criteria:

Adults (non-pregnant) with sound judgment

Chronic TMJ pain lasting at least 12 months

Documented failure of at least two previous treatment modalities

Exclusion Criteria:

Failure to meet inclusion criteria

Missing at least two follow-up visits within the specified timeframe

Data Handling and Confidentiality:

All data will be anonymized and stored in a secure, password-protected Excel file within the department. Only approved researchers will have access. Patient identifiers will be replaced with study codes. No personal identifying information will be published or disclosed.

Ethical Considerations:

The study will only begin after approval by the institutional Helsinki (ethics) committee. All participants will provide written informed consent after receiving a thorough explanation of the study. Participation is voluntary and will not impact the quality or accessibility of their medical care. Patients may withdraw at any time without consequence.

Statistical Analysis:

The main outcomes (VAS scores, analgesic use, and mouth opening) will be compared before and after treatment using standard statistical methods. Subgroup analyses will explore correlations between outcomes and demographic/clinical variables such as age, sex, and previous treatment history.

ELIGIBILITY:
Inclusion Criteria:

* Adults (non-pregnant) with sound judgment
* Chronic TMJ pain lasting at least 12 months
* Documented failure of at least two previous treatment modalities

Exclusion Criteria:

* not meeting inclusion criteria
* Missing at least two follow-up visits within the specified timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic temporomandibular joint (TMJ) pain who attend the TMJ clinic at Beni Zion hospital, part of the Department of Oral and Maxillofacial Surgery. Participants are individuals who have experienced TMJ-related pain for at least one year and have not responded adequately to at least two prior treatment modalities (e.g., physiotherapy, medications, splints, or alternative therapies). Eligible patients will be those for whom a peripheral nerve block has been selected as part of their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
VAS pain intensity | One year
  Pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable), before and after treatment.

SECONDARY OUTCOMES:
Mouth opening meausurement | One year
  Maximal mouth opening (in millimeters) will be measured before and after treatment.
Change in analgesic use | One year
  Patient-reported use of pain medications before and after the nerve block treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Haifa, North, Israel